CLINICAL TRIAL: NCT06823297
Title: Can Neoadjuvant Chemoradiotherapy be Omitted in cT2N+ and cT3 Mid-rectal Cancer: A Prospective, Observational Cohort Study
Brief Title: Can Neoadjuvant Chemoradiotherapy be Ommited in Mid-rectal Cancer
Acronym: CANO
Status: Not yet recruiting | Type: Observational
Sponsor: Turkish Society of Colon and Rectal Surgery (Other)
Collaborators: Baskent University (Other); Dokuz Eylul University (Other); Halic University (Other); Acibadem Kent Hospital (Other); Istanbul Health and Technology University (Other)
Responsible Party: Sponsor
Other Study IDs: KA24/461
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Mid-Rectal Cancer; Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: Mid-Rectal Cancer; Radiotherapy; Mesorectal fascia
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Upfront TME group: Patients who underwent surgery without receiving neoadjuvant chemoradiotherapy
  Interventions: Other: Total mesorectal excision
- Neoadjuvant chemoradiotherapy group: Patients who received neoadjuvant chemoradiotherapy before surgery
  Interventions: Other: Neoadjuvant Chemotherapy followed by total mesorectal excision

INTERVENTIONS:
Other: Total mesorectal excision — Direct surgery without receiving neoadjuvant chemoradiotherapy
  Groups: Upfront TME group
Other: Neoadjuvant Chemotherapy followed by total mesorectal excision — Neoadjuvant chemoradiotherapy treatment regimens (including conventional chemoradiotherapy/radiotherapy/chemotherapy regimens or total neoadjuvant chemoradiotherapy regimens) before surgery
  Groups: Neoadjuvant chemoradiotherapy group

SUMMARY:
This project aims to compare the oncological and functional outcomes of patients with mid-rectal cancer who have a low risk of local recurrence (without MRF involvement) and who either receive or do not receive neoadjuvant chemoradiotherapy (nCRT).

Main Question:

H0: In mid-rectal cancer patients without MRF involvement (cT2N+ and cT3Nx), there is no difference in 3-year disease-free survival between direct TME and TME after nCRT.

H1: In mid-rectal cancer patients without MRF involvement (cT2N+ and cT3Nx), direct TME is associated with worse 3-year disease-free survival compared to TME after nCRT.

Participants already taking both interventions as part of their regular medical care for rectal cancer will be recruited in a prospective database for 5 years.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (nCRT) followed by total mesorectal excision (TME) is the standard treatment for patients with locally advanced rectal cancer. This approach has been shown to improve local control and reduce recurrence rates. However, there is no clear evidence showing the advantage of neoadjuvant CRT in high and middle rectal tumors without involvement of mesorectal fascia (MRF). The MERCURY study demonstrated that preoperative MRI-predicted positive CRM is an independent factor for local recurrence. Following this study, the selective use of nCRT in patients at high risk of local recurrence has been proposed.

The ESMO guidelines indicate that T3a/b rectal tumors located above the levator muscles, without involvement of the circumferential resection margin (CRM) or extramural venous invasion (EMVI), are associated with a very low risk of local recurrence. Consequently, they suggest that upfront TME may be an appropriate treatment option for this subgroup of patients. This recommendation remains unchanged in the presence of lymph node involvement within the same group. For clinically staged cT3a/b mid- or high-rectal tumors with clear CRM and no evidence of EMVI, the routine use of nCRT remains a subject of debate. If the surgeon consistently performs high-quality total mesorectal excision (TME), upfront surgery may be a suitable treatment option for this subgroup of patients.

In line with these recommendations, some surgeons perform upfront TME for patients with T2-3 node-positive mid-rectal cancer in the absence of MRF involvement. However, in these cases, the common approach is to administer neoadjuvant chemoradiotherapy. This study seeks to observe whether upfront TME achieves similar 3-year disease-free survival compared to the standard approach of nCRT followed by TME in patients with cT2N+ and cT3Nx mid-rectal cancer without mesorectal fascia involvement.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed rectal cancer
* Rectal cancer within 6-12 cm from anal verge confirmed by sigmoidoscopy or located between the anorectal junction and peritoneal reflection identified by MRI
* Clinical local staging performed by MRI
* cT2N+, cT3N0 and cT3N+ tumors
* Patients without mesorectal fascia involvement assessed by MRI (≤1 mm)
* Patients without pathological (short axis ≥7 mm) lateral (extramesorectal) lymph nodes on MRI
* Patients without EMVI on MRI

Exclusion Criteria:

* cT4 tumors
* Stage IV disease
* Patients with MSI (+) in TME pathology
* PAtients who received neoadjuvant immunotherapy
* Emergency surgery
* Clinical obstruction
* Previous pelvic radiotherapy
* Patients treated without a multidisciplinary council decision
* Inflammatory bowel diseases (Crohn's disease, Ulcerative colitis)
* Familial adenomatous polyposis (FAP), attenuated FAP, and other polyposis syndromes
* Hereditary non-polyposis colorectal cancer (Lynch syndrome)
* Synchronous colon tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven rectal cancer patients with locally advanced disease (cT2N0-T3N0-N+), but without distant metastases or high-risk features such as mesorectal fascia involvement, lateral nodes, EMVI or adjacent organ invasion (cT4).
Sampling Method: Probability Sample
Enrollment: 436 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2035-08-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  The proportion of patients who remain free of disease recurrence (local or distant) three years after surgical intervention. DFS will be assessed through clinical evaluations, imaging studies, and pathology reports at regular follow-up intervals.

SECONDARY OUTCOMES:
Overall Survival | 3 and 5 years
  The proportion of patients alive at 3 and 5 years post-treatment, regardless of disease status.
Local Recurrence Rate | 3 years and 5 years
  The percentage of patients experiencing tumor recurrence at the primary site (anastomosis or pelvis) within 3 and 5 years.
Colorectal Cancer Specific Quality of Life | Baseline, 1 year, 3 years and 5 years
  Patient-reported outcomes assessed using the New Cleveland Clinic Colorectal Cancer Quality of Life Questionnaire
Bowel Dysfunction Related Quality of Life | Baseline, 1 year, 3 years and 5 years
  Patient-reported outcomes assessed using the low-anterior resection syndrome (LARS) score.

CONTACTS AND LOCATIONS:
Overall Officials: Feza Karakayali, Prof., Study Chair — Baskent University; Aras Emre Canda, Prof., Principal Investigator — Acibadem Kent Hospital; Ilknur Erenler Bayraktar, Prof., Principal Investigator — Halic University; Onur Bayraktar, Prof., Principal Investigator — Memorial Sisli Hospital; Cigdem N Arslan, Prof., Study Director — Istanbul Health and Technology University; Tayfun Bisgin, Prof., Principal Investigator — Dokuz Eylul University
Locations (5):
- Turkey (Türkiye) (5):
  - Baskent University, Ankara
  - Istanbul Health and Technology University, Istanbul
  - Memorial sisli Hospital, Istanbul
  - Acibadem Kent Hospital, Izmir
  - Dokuz Eylul University, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Yes, we plan to share de-identified individual participant data (IPD) related to primary and secondary outcomes. The data will be available to qualified researchers upon reasonable request, starting 6 months after publication of the study results and for up to 5 years. Data will be shared via a secure data repository, and access will require an approved data-sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months to 5 years
URL: https://arastirma.tkrcd.org.tr/

REFERENCES:
- [Background] Patel UB, Taylor F, Blomqvist L, George C, Evans H, Tekkis P, Quirke P, Sebag-Montefiore D, Moran B, Heald R, Guthrie A, Bees N, Swift I, Pennert K, Brown G. Magnetic resonance imaging-detected tumor response for locally advanced rectal cancer predicts survival outcomes: MERCURY experience. J Clin Oncol. 2011 Oct 1;29(28):3753-60. doi: 10.1200/JCO.2011.34.9068. Epub 2011 Aug 29. PMID 21876084
- [Background] Ruppert R, Kube R, Strassburg J, Lewin A, Baral J, Maurer CA, Sauer J, Junginger T, Hermanek P, Merkel S; other members of the OCUM Group. Avoidance of Overtreatment of Rectal Cancer by Selective Chemoradiotherapy: Results of the Optimized Surgery and MRI-Based Multimodal Therapy Trial. J Am Coll Surg. 2020 Oct;231(4):413-425.e2. doi: 10.1016/j.jamcollsurg.2020.06.023. Epub 2020 Jul 19. PMID 32697965
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Derived] Karakayali F, Arslan C, Bisgin T, Erenler Bayraktar I, Bayraktar O, Canda AE. Can neoadjuvant chemoradiotherapy be omitted in cT2N+ and cT3 mid-rectal cancer: Protocol for a prospective, observational, cohort study (CANO). PLoS One. 2025 Nov 5;20(11):e0321819. doi: 10.1371/journal.pone.0321819. eCollection 2025. PMID 41191581